CLINICAL TRIAL: NCT02461329
Title: Comparison of the Effects of Gelatine (Gelofusine ® B. Braun) Versus Crystalloid Solution (Ringerfundin ® B. Braun) for Volume Therapy on Coagulation, Thrombocyte Function and Thrombelastometry (ROTEM ®), in Elective Hip Replacement Surgery
Brief Title: Comparison of the Effects of Gelatine Versus Balanced Crystalloid Solution for Volume Therapy
Acronym: Gelaring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kratochvil Milan, MD (Other)
Collaborators: IBA - Masaryk University Institute of biostatistics and analyses (Unknown)
Responsible Party: Sponsor-Investigator, Kratochvil Milan, MD, Research coordinator, Brno University Hospital
Organization: Brno University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FN-Brno
Record Dates: First submitted 2015-04-16; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hemorrhage, Surgical; Hip Replacement, Total; Thrombocytopathy
Keywords: Hip Replacement, Total; Gelatine solution; Balanced Crystaloid Solution; Volume therapy; Platelet aggregation
MeSH Terms: conditions — Blood Loss, Surgical; Blood Platelet Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelatine solution (Experimental): Gelofusine will be administrated like "fluid challenge" - 250ml of solution will be infused within 5 minutes in case of hypotension ( mean arterial pressure - MAP below 65 mmHg or below 70mmHg in patient with chronic hypertension disease).
  The blood pressure and heart rate before and after fluid challenge will be recorded.
  Interventions: Drug: Gelofusine® B. Braun
- Balanced Crystaloid solution (Experimental): Ringerfundin will be administrated like "fluid challenge" - 250ml of solution will be infused within 5 minutes in case of hypotension ( mean arterial pressure - MAP below 65 mmHg or below 70mmHg in patient with chronic hypertension disease).
  The blood pressure and heart rate before and after fluid challenge will be recorded.
  Interventions: Drug: Ringerfundin ® B. Braun

INTERVENTIONS:
Drug: Gelofusine® B. Braun — Volume therapy by Gelatine solution infusion via intravenous boluses to achieve hemodynamic targets
  Arms: Gelatine solution
Drug: Ringerfundin ® B. Braun — Volume therapy by Balanced Crystaloid solution solution infusion via intravenous boluses to achieve hemodynamic targets
  Arms: Balanced Crystaloid solution

SUMMARY:
The purpose of the study is to determine whether volume therapy with a solution of gelatine has negative impact on coagulation, platelet function, renal function in comparison with crystaloid solution (Ringerfundin).

DETAILED DESCRIPTION:
After obtaining the research ethics committee approval, 50 patients, undergoing elective surgery for hip replacement will be included. The informed consent must be signed prior to randomization. After arriving to the operation theatre, the patients informed consent and inclusion and exclusion criteria will be reviewed. Afterwards, the patients will be randomized in one of two groups. Prior to the anaesthesia induction, blood for the thrombocyte function test, coagulation tests and thrombelastometry wil be drawn via a metal cannula. A large bore peripheral venous cannula (G18 or more) will be introduced. In case of a ASA status of III and higher based on cardiovascular morbidity an arterial catheter via the radial artery for invasive blood pressure monitoring will be introduced. Urinary catheter will be introduced to monitor intraoperative diuresis. A continuous crystalloid infusion n a dose of 5 ml/kg/hour will be administered for basal fluid substitution. The volume replacement using blinded gelatine/crystalloid solution will be performed via fluid challenge (repeated 250 ml fluid boluses during a 5 minute interval) to hemodynamic targets (increase in blood pressure, decrease in heart rate), in case of a decrease of MAP to 65 mm Hg (16) or to 70 mmHg in preexisting hypertension. The hemodynamic variables before and after fluid challenge will be exactly recorded. In case the patient hemodynamics does dot respond to a fluid challenge, or in case of a drop of blood pressure to less than 55 mmHg, a bolus of 5-10 mg of ephedrine (repeatedly) will be administered. Further recorded variables will be: blood loss (suctioning, sponges), diuresis, number of transfusions administered. Repetitive hemoglobin concentration tests using the HemoCue 201+ device will be performed and an intraoperative blood transfusion trigger of 90 g/l of hemoglobin concentration will be used, 100 g/l in case of a patient with chronic cardiovascular or respiratory disease (5). After reaching the blood loss of 1000 ml, blood samples will be drawn for laboratory hemoglobin concentration and coagulation testing. The trigger for platelet transfusion will be a thrombocyte count of less than 50000 x 109, or sings of platelet dysfunction on thrombelastometry. Tranexamic acid will be administered in case of signs of fibrinolysis on thrombelastometry or in case of life threatening bleeding. At the end of surgery, a second blood sample for platelet function test, thrombelastometry, full blood count and standard coagulation tests will be drawn. The amount of blinded study infusion, continuous crystalloid solution, transfusions and ephedrine administered, diuresis and blood loss will be recorded. Blood urea and creatinine, diuresis, coagulations and full blood count will be recorded postoperatively. Hospital and ICU length of stay, hospital and 90-day mortality will be followed.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for elective hip replacement surgery
* age between 19-85 years
* signed informed consent

Exclusion Criteria:

* informed consent not signed
* traumatic hip fracture
* anemia (hemoglobin level < 100 g/l)
* allergy to study drug and/or multiple allergies
* chronic heart failure with LVEF < 30%
* shock states
* coagulopathy
* thrombocytopenia
* thrombocytopathy
* chronic kidney disease with oliguria
* chronic antiplatelet drug medications

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of coagulation status and platelet function | perioperative, an expected average of 2 hours
  Before and after the surgery (in OR) the investigator will obtain a blood sample from subject, standard coagulation test will be performed (INR, PT, aPTT, thrombin time), the investigator will perform ROTEM tests: EXTEM, INTEM and FIBTEM assay and blood sample will be tested for thrombocyte function - aggregation with ADP, collagen, epinephrine, TRAP - thrombin receptor-activated peptide.

SECONDARY OUTCOMES:
Blood loss | perioperative, an expected average of 2 hours
  Amount of blood loss during the surgery and in the postoperative period
Renal function | 2 days after surgery
  serum creatinine and blood urea nitrogen will be recorded 48 hours after surgery
Transfusion needs | hospital stay, an expected average of 1 week
  Number of transfusion units administered during whole hospital stay

OTHER OUTCOMES:
Perioperative complications | hospital stay, an expected average of 1 week
  Investigators will review all records after patient dismission and search for any complications related to medical care

CONTACTS AND LOCATIONS:
Overall Officials: Milan Kratochvil, MD, Principal Investigator — FN Brno; Milan Kratochvil, MD, Study Director — FN Brno; Roman Gál, Prof, MD, Ph.D, Study Chair — Fn Brno